CLINICAL TRIAL: NCT03318458
Title: Effects of a Program of Pilates Exercises in Spanish Women With Fibromyalgia
Brief Title: Pilates Exercises in Spanish Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Physiotherapy, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Jaen University
Record Dates: First submitted 2017-10-03; First posted 2017-10-24 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Fall Due to Loss of Equilibrium
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
  All measurements given above will be made both to the control group and to the experimental group just prior to the start of the intervention, and immediately after and six months after the end of this period, and the results will be recorded in a data record
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental)
  Interventions: Other: Pilates
- No intervention group (No Intervention)

INTERVENTIONS:
Other: Pilates — The duration of the intervention is 12 weeks, with 2 sessions per week of Pilates. Each session lasts approximately 1 hour and is structured in three parts: initial warm-up, which reviews the basic principles of the Pilates Method (centralization, concentration, movement control, breathing, movement precision and fluency) of 10 minutes duration, a 40-45 minute Pilates session and finally 10 minutes of guided relaxation. No complement was used (magic rings, fitball, elastic bands, etc.) during classes
  Arms: Pilates group

SUMMARY:
To analyze the effects of a Pilates exercise program in Spanish postmenopausal women with Fibromyalgia

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (Control group and experimental group), in which a pre-treatment-postest design has been used.

The study will define two groups:

* A control group (CG) that will not be submitted to treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity and will be given a guide to recommendations for promoting physical activity.
* An experimental group (GE) that after an initial evaluation will undergo a physical training program based on Pilates exercises.

Once the intervention is finished, it will be submitted to a final evaluation to see if there is a difference or not with the results obtained at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* No menstrual activity for at least 12 months.
* Present Fibromyalgia.
* Do not participate in a weight loss program.
* Be able to understand the instructions, programs and protocols of this project.

Exclusion Criteria:

* Contraindications for conducting physical tests.
* Diseases that limit the static and dynamic balance and physical activity. -
* Central or peripheral vestibular or nerve alterations.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Dynamometer | At the beginning and at three months
  Dynamometer will be employed to assess hand grip stregth
ABC-16 (Activities Specific Balance Confidence Scale) | At the beginning and at three months
  Questionnaire that assesses balance confidence in performing activities of daily living. It is calculated by adding up the 16 responses of the questionnaire, with 0 being the minimum score and 100 being the maximum score. The higher value represents a better result.
FES-I (Falls Efficacy Scale-International) | At the beginning and at three months
  Questionnaire that evaluates the fear of falling. It is calculated by adding up all the answers in the questionnaire, 16 being the minimum score and 64 the maximum score. The higher value represents a worse result.
FSS (Fatigue Severity Scale) | At the beginning and at three months
  A self-report scale describing the severity of fatigue and the impact of fatigue on activities of daily living. It is calculated by adding up the 9 answers of the questionnaire, being 9 the minimum score and 63 the maximum score. The higher value represents a worse result.
FIQ (Fybromialgia Impact Questionnaire) | At the beginning and at three months
  A questionnarie that evaluates the impact of fibromyalgia on the patient's quality of life.The total score is the addition of the scores of all its sections. In the case that there were left some unanswered, all the other ones are added up and the score is divided by the number of items answered and multiplied by 10, with the result that the final score of the FIQ is from 0 to 100. A higher score means a greater impact of the disease on the patient.
VAS-Fatigue | At the beginning and at three months
  Fatigue assessed by a Visual Analogue Scale (10 cm). The patient marks the intensity of the fatigue on a numerical scale of 0-10, with 0 being the minimum score and 10 being the maximum score. The higher value represents a worse result.
VAS-pain | At the beginning and at three months
  Pain assessed by a Visual Analogue Scale (10 cm). The patient on a numerical scale of 0-10 marks the intensity of the pain, with 0 being the minimum score and 10 the maximum score. The higher value represents a worse result.
PSQI (Pittsburgh Sleep Quality Index) | At the beginning and at three months
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result.
HADS (The Hospital Anxiety And Depression) | At the beginning and at three months
  A reliable, valid and practical screening tool for identifying and quantifying anxiety and/or depression in non- patients. It is calculated by the sum of the 14 questions in the questionnaire divided into two subscales: anxiety (questions 1, 3, 5, 7, 9, 11, 13) and depression (questions 2, 4, 6, 8, 10, 12, 14). The higher value represents a worse result.
SF-36 (The Short Form-36 Health Survey) | At the beginning and at three months
  Used extensively for assessing health-related quality of life. It is calculated by adding the 36 questionnaires divided into 9 subscales: general health, health change, physical function, physical role, role or emotional performance, social function, physical or body pain, vitality and mental health. Each item is rated 0-1-2-3-4 points with 0 being the best score.
INBODY | At the beginning and at three months
  Valid and reliable tool to quantify and measure the 4 major components of body composition: Water, Protein, Minerals and Fat
Bone Mineral Content (BMC) | At the beginning and at three months
  Is mineral mass in bone
Body Weight: is the sum of Body Fat and Fat Free Mass. | At the beginning and at three months
  Is the sum of Body Fat and Fat Free Mass
Skeletal Muscle Mass (kg) | At the beginning and at three months
  Is computed based on muscle mass of the limbs, which is almost composed of skeletal muscle and takes up about 70% of total body skeletal muscle
Lean Body Mass | At the beginning and at three months
  The amount of lean body mass
Body Fat Mass | At the beginning and at three months
  The standard range of Body Fat Mass is ascertained by calculating an examinee Body Fat Mass as compared to the standard weight and standard Body Fat Mass
Percent of Body Fat (%) | At the beginning and at three months
  Indicates the percentage of body fat to body weight
BMI (Body Mass Index) | At the beginning and at three months
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat
Segmental Analysis | At the beginning and at three months
  Is the technology that assumes the body as five cylinders of four limbs and trunk and measures the impedance of these parts separately. Segmental body composition analysis provides segmental measurement of body water, muscle mass, and fat free mass
TUG (Timed Up and Go test) | At the beginning and at three months
  Is a simple test used to assess a person's mobility and physical function
CT10P | At the beginning and at three months
  Test that evaluates the balance by walking along a straight line
MRS (Menopause Rating Scale) | At the beginning and at three months
  assesses the severity of menopause-related complaints and the impact on health-related quality of life. Calculated by adding up the 11 questions in the questionnaire. Each item has a score of 0-1-2-3-4, with 4 being the worst score.
STABILOMETRIC PLATFORM | At the beginning and at three months
  instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions
X mean | At the beginning and at three months
  Mean value of the lateral oscillations of the Pressure Center
Y mean | At the beginning and at three months
  Mean value of the anteroposterior oscillations of the Pressure Center
RMS X | At the beginning and at three months
  Mean position of the center of pressure in the mediolateral plane
Length | At the beginning and at three months
  Length of the path described by the center of pressure
Area | At the beginning and at three months
  Area of the path described by the center of pressure
Velocity | At the beginning and at three months
  Is an estimate of the average velocity of displacement of the center of pressures of the subject during the whole test
Chair Sit and Reach Test | At the beginning and at three months
  To test low back and hamstring flexibility
Back Scratch Test | At the beginning and at three months
  To measure general shoulder range of motion
30-Second Chair Stand Test | At the beginning and at three months
  To test leg strength and endurance
Height | At the beginning and at three months
  The distance between the lowest and highest points of a person standing upright
Wais Circumference | At the beginning and at three months
  Is used to assess central fat distribution and degree of abdominal obesity
Hip Circumference | At the beginning and at three months
  It is the greatest circumference of hip
Waist-To-Hip Ratio | At the beginning and at three months
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement

CONTACTS AND LOCATIONS:
Locations (1):
- AFIXA, Jaén, Spain